## STATISTICAL ANALYSIS PLAN

# Delayed loading following repair of ruptured Achilles tendon — A randomized controlled trial

# Index:

| INDEX: | 2 |
|---------------------------|---|
| BACKGROUND | 3 |
| Purpose | 3 |
| Hypotheses | |
| STUDY DESIGN | 3 |
| Participants | |
| Blinding | |
| Sample size calculation | |
| OUTCOME ASSESSMENTS | 5 |
| Primary outcome | |
| Secondary outcomes | |
| POPULATION TO BE ANALYZED | 5 |
| Intension-to-treat (ITT) | ε |
| Per protocol (PP) | |
| ANALYSIS | 6 |
| Primary outcome | |
| Secondary outcome | |
| Table of the analysis | |
| REFERENCES | |

## Background

Leisure time physical activity is unquestionably associated with numerous health benefits. However, some of these recreational activities are also accompanied with some increased risk of injury. For example, there appears to be an increased risk of Achilles tendon ruptures with some recreational sports (1). Specifically, this increased incidence can be seen in high-impact sports, including badminton, volleyball, and soccer (2, 3). Acute Achilles tendon ruptures occurs in both men and women but is most frequent in men 30-50 years of age that participate in recreational sports periodically (1, 4, 5). The prevalence is reported to be ~ 18 per 100,000 per year, and the incidence appear to be on the rise (1, 4-6). Yet, evidenced based knowledge of how to best rehabilitate the injury after repair of the rupture is largely absent in the literature, which likely contributes to the reports of persistent muscle weakness, tendon elongation and incomplete return to pre-injury level (7-18). It has been suggested that preventing tendon elongation during rehabilitation improves the clinical outcome, which is the very aim of this project.

#### Purpose

The purpose of the present study is to investigate if delayed loading following surgical treated Achilles tendon rupture influence the clinical outcome and muscle and tendon structure after one year.

## Hypotheses

We hypothesize that delaying the gradual introduction of loading in the initial 26 weeks may reduce the heel-rise deficit (primary outcome) and thus improve the clinical outcome one year after surgery (primary endpoint).

# Study design

This study is a single-blinded prospective randomized controlled superiority trial with 2 parallel arms. (The study will be registered by ClinicalTrials.gov). We will examine if delaying initiation of loading in the initial 26 weeks will influence the tendon healing and elongation compared to current accepted clinical guidelines for rehabilitation ('accelerated rehabilitation') of surgically repaired Achilles tendon ruptures. One arm will include current clinical practice that calls for partial weight bearing from week 3, full weight bearing from week 7, and total bracing time 6

weeks. The other arm will not be allowed partial weight bearing with the use of crutches until week 7 and full weight bearing until week 13, and total bracing time is 12 weeks.

#### **Participants**

The patient recruitment will be achieved in-house from the emergency clinic and the orthopedic surgery department at Bispebjerg and Frederiksberg Hospital. Potential participants are either identified by the diagnosing doctor, or by the primary investigator through screening of the orthopedic surgery-lists. Furthermore, features of the SP-journal system will be used to support recruitment. For patients identified by the diagnosing doctor, once the diagnosis of Achilles tendon rupture is established, patients are orally informed about the study and if interested in participating they will receive the written attending information ("Deltagerinformation"). Patients identified through the orthopedic surgery-lists will be approached by the primary investigator in person on the day of surgery and will be given the same oral and written information as those identified by the diagnosing doctor. Patients interested in participating will either contact the primary investigator or will be approached in person on the day of surgery, to be screened for eligibility. The orthopedic surgeons will assess all patients after standard procedures and, if surgical intervention is decided, patients will undergo the standard surgical procedure. After surgery, patients will be randomized to one of the two rehabilitation groups:

- A) Early mobilization. This constitutes the currently accepted regime and is therefore considered the control group.
- B) Delayed mobilization.

Randomization procedure is performed using a computer-generated block randomization (blocks of 4) procedure.

#### Blinding

Because this is an "open-label" trial the health professionals delivering the interventions and the participants will not be blinded to treatment allocation. Outcome assessors will be blinded to treatment allocation whenever possible: This is of outmost importance, and participants are requested not to disclose their allocation when outcomes are assessed.

#### Sample size calculation

Based on heel-rise deficit (primary outcome) relative to the uninjured side ( $u_A$ =76 %,  $u_B$ =90 %,  $\sigma$ =16) a sample of n=21 is required to detect a difference with a power of 80% (19). To account for drop-outs a sample of 24 in each arm will be recruited.

#### Outcome assessments

#### Primary outcome

The primary outcome is heel-rise height deficit on the injured side relative to the uninjured side at one-year follow-up.

#### Secondary outcomes

The following outcomes are assessed as secondary outcomes:

- Heel-rise work.
- Achilles Tendon Total Rupture Score (ATRS).
- Gastrocnemius and soleus muscle fascicle length and pennation angle.
- Gastrocnemius and soleus tendon and lower limb muscle cross-sectional area.
- Plantarflexion Isokinetic muscle strength.
- Physical actively level (PAS).
- Tendon length.
- Achilles Tendon Resting Angle (ATRA).

# Population to be analyzed

To be included in the study, participants must meet the following in- and exclusion criteria:

#### **Inclusion criteria**

- Diagnosed with a traumatic, complete mid-substance Achilles tendon rupture
- No contraindications for MRI
- Presented within 14 days from injury
- Adult (18 to 60 years)
- Understand Danish
- Manage transport to/from the hospital on their own

#### **Exclusion criteria**

- Other injuries affecting their lower limb functions
- Prior Achilles tendon rupture
- Re-rupture
- Smoking
- Systemic diseases influencing tendon healing
- Anticoagulation treatment
- Inability to follow rehabilitation or complete follow-ups
- Immunosuppressive treatment including systemic corticosteroid treatment.

#### Intension-to-treat (ITT)

All participants who are randomized.

#### Per protocol (PP)

All participants who adhere to the major criteria in the protocol and completed the whole study period and attended 1 year follow-up. Participants with missing data on any of the variables in the model will be excluded from the specific analysis at the specific timepoint.

## **Analysis**

All outcomes will be reported using descriptive statistics. Normally distributed data by the mean and standard deviation and skewed distributions by the median and interquartile range. Binary and categorical variables will be presented using counts and percentages. SAS and Prism will be used for all statistical analysis. Analyses in addition to the descriptive statistics are described below.

#### Primary outcome

The primary analysis will be an assessment of the between group difference in heel-rise height deficit on the injured side relative to the uninjured side ((uninjured-injured/uninjured) x 100)) at one-year follow-up. Intention-to-treat and per-protocol analysis will be conducted. The criteria for being included in the per-protocol analysis is having attended 1 year follow-up tests. An unpaired students t-test will be used to analyze the primary outcome (heel-rise deficit) at the primary endpoint (one year).

#### Secondary outcome

A mixed model (group x time) that includes all timepoints will be used to analyze the secondary outcomes and the primary outcome. In addition, a correlation matrix for the changes in secondary and primary outcome will be performed, followed by a multiple regression. ATRA will be compared with MRI and correlated.

#### Table of the analysis

| OUTCOME | TIMEPOINTS | UNPAIRED<br>T-TEST | MIXED MODEL | CORRELATION | MULTIPLE<br>REGRESSION |
|---|---|---|---|---|---|
| MRI | 4 | | х | Х | х |
| Tendon length | | | | | |
| CSA tendon | | | | | |
| CSA muscle | | | | | |
| Free fat fraction | | | | | |
| ULTRASOUND | 4 | | х | Х | Х |
| Fascicle length | | | | | |
| Pennation angle | | | | | |
| Thickness muscle | | | | | |
| Doppler tendon | | | | | |
| Thickness tendon | | | | | |
| HEELRISE | 2 | | X | Х | Х |
| Work | | | | | |
| Hight | | | | | |
| Repetitions | | | | | |
| ATRA | 2 | | х | х | х |
| MUSCLE STRENGTH | 1 | x | | x | х |
| ATRS | 2 | X | | Х | Х |
| PAS | 2 | X | | Х | Х |
| LIKERT SCALE | 1 | X | | | |

### References

- 1. Houshian S, Tscherning T, Riegels-Nielsen P. The epidemiology of Achilles tendon rupture in a Danish county. Injury. 1998;29(9):651-4.
- 2. Huttunen TT, Kannus P, Rolf C, Fellander-Tsai L, Mattila VM. Acute achilles tendon ruptures: incidence of injury and surgery in Sweden between 2001 and 2012. The American journal of sports medicine. 2014;42(10):2419-23.
- 3. Kujala UM, Sarna S, Kaprio J. Cumulative incidence of achilles tendon rupture and tendinopathy in male former elite athletes. Clinical journal of sport medicine: official journal of the Canadian Academy of Sport Medicine. 2005;15(3):133-5.
- 4. Nillius SA, Nilsson BE, Westlin NE. The incidence of Achilles tendon rupture. Acta Orthop Scand. 1976;47(1):118-21.
- 5. Maffulli N, Waterston SW, Squair J, Reaper J, Douglas AS. Changing incidence of Achilles tendon rupture in Scotland: a 15-year study. Clin J Sport Med. 1999;9(3):157-60.
- 6. Leppilahti J, Puranen J, Orava S. Incidence of Achilles tendon rupture. Acta Orthop Scand. 1996;67(3):277-9.
- 7. Moller M, Lind K, Movin T, Karlsson J. Calf muscle function after Achilles tendon rupture. A prospective, randomised study comparing surgical and non-surgical treatment. Scand J Med Sci Sports. 2002;12(1):9-16.
- 8. Suchak AA, Spooner C, Reid DC, Jomha NM. Postoperative rehabilitation protocols for Achilles tendon ruptures: a meta-analysis. Clin Orthop Relat Res. 2006;445:216-21.
- 9. Khan RJ, Fick D, Keogh A, Crawford J, Brammar T, Parker M. Treatment of acute achilles tendon ruptures. A meta-analysis of randomized, controlled trials. J Bone Joint Surg Am. 2005;87(10):2202-10.
- 10. Mullaney MJ, McHugh MP, Tyler TF, Nicholas SJ, Lee SJ. Weakness in end-range plantar flexion after Achilles tendon repair. Am J Sports Med. 2006;34(7):1120-5.
- 11. Amin NH, Old AB, Tabb LP, Garg R, Toossi N, Cerynik DL. Performance Outcomes After Repair of Complete Achilles Tendon Ruptures in National Basketball Association Players. Am J Sports Med. 2013.
- 12. Silbernagel KG, Steele R, Manal K. Deficits in heel-rise height and achilles tendon elongation occur in patients recovering from an Achilles tendon rupture. Am J Sports Med. 2012;40(7):1564-71.
- 13. Silbernagel KG, Nilsson-Helander K, Thomee R, Eriksson BI, Karlsson J. A new measurement of heel-rise endurance with the ability to detect functional deficits in patients with Achilles tendon rupture. Knee surgery, sports traumatology, arthroscopy: official journal of the ESSKA. 2010;18(2):258-64.
- 14. Olsson N, Nilsson-Helander K, Karlsson J, Eriksson BI, Thomee R, Faxen E, et al. Major functional deficits persist 2 years after acute Achilles tendon rupture. Knee Surg Sports Traumatol Arthrosc. 2011.
- 15. Barfod KW, Sveen TM, Ganestam A, Ebskov LB, Troelsen A. Severe Functional Debilitations After Complications Associated With Acute Achilles Tendon Rupture With 9 Years of Follow-Up. J Foot Ankle Surg. 2017.
- 16. Heikkinen J, Lantto I, Flinkkila T, Ohtonen P, Niinimaki J, Siira P, et al. Soleus Atrophy Is Common After the Nonsurgical Treatment of Acute Achilles Tendon Ruptures: A Randomized Clinical Trial Comparing Surgical and Nonsurgical Functional Treatments. Am J Sports Med. 2017;45(6):1395-404.
- 17. Lantto I, Heikkinen J, Flinkkila T, Ohtonen P, Kangas J, Siira P, et al. Early functional treatment versus cast immobilization in tension after achilles rupture repair: results of a prospective randomized trial with 10 or more years of follow-up. The American journal of sports medicine. 2015;43(9):2302-9.
- 18. Rosso C, Buckland DM, Polzer C, Sadoghi P, Schuh R, Weisskopf L, et al. Long-term biomechanical outcomes after Achilles tendon ruptures. Knee Surg Sports Traumatol Arthrosc. 2015;23(3):890-8.
- 19. Eliasson P, Agergaard AS, Couppe C, Svensson R, Hoeffner R, Warming S, et al. The Ruptured Achilles Tendon Elongates for 6 Months After Surgical Repair Regardless of Early or Late Weightbearing in Combination With Ankle Mobilization: A Randomized Clinical Trial. The American journal of sports medicine. 2018;46(10):2492-502.